CLINICAL TRIAL: NCT02857543
Title: Plant-Based, No-Added-Fat or American Heart Association or Mediterranean Diets a Prospective Randomized Trial: Impact on Cardiovascular Risk in Obese Children With Hypercholesterolemia and in One of Their Parents
Brief Title: Plant-Based, American Heart Assoc. or Mediterranean Diets In 9-18 yo With BMI >95%, Cholesterol >169 and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, michael macknin, Professor of Pediatrics, Cleveland Clinic Lerner College of Medicine of CWRU, Cleveland Clinic, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-745
Record Dates: First submitted 2016-07-01; First posted 2016-08-05 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Obesity; Hypercholesterolemia; Cardiovascular Disease
MeSH Terms: conditions — Obesity; Hypercholesterolemia; Cardiovascular Diseases | interventions — Diet, Plant-Based; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- plant-based diet (Active Comparator): Plant-based diet with as few added oils and fats as possible
  Interventions: Other: Plant-Based Diet
- American Heart Association (Active Comparator): Diet encourages fruits, vegetables, whole grains, and low sodium intake but permits non-whole grains, low-fat dairy, selected plant oils, and lean meat and fish in moderation.
  Interventions: Other: American Heart Association Diet
- Mediterranean (Active Comparator): Diet encourages fruits, vegetables, whole grains, and low sodium intake but permits non-whole grains, low-fat dairy, selected plant oils, with more emphasis on fish and extra virgin olive oil and/or nuts.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Plant-Based Diet
  Arms: plant-based diet
Other: American Heart Association Diet
  Arms: American Heart Association
Other: Mediterranean Diet
  Arms: Mediterranean

SUMMARY:
The purpose of this research is to investigate the effects of a PB no- added-fat and the AHA and MED in obese (BMI >95%) children ages 9-18 with hypercholesterolemia (>169 mg/dl) and a parent or guardian. Eligible patients will be identified by utilizing the Pediatric Obesity Registry. When possible, in-person discussions or phone calls with their primary or tertiary care physicians will introduce eligible patients and their parents to the study. All eligible patients and parents will receive letters describing the study and requesting their participation. Subjects can choose not to participate in the study, and their health care will not be affected in any way. Subjects not participating will be asked if they are willing to answer a brief questionnaire about why they chose not to participate. The proposed study will be carried out for a total of 52 weeks. The investigators expect to recruit a total of 180 participants (30 children and 30 parents/guardians in each of the three groups). Each child and parent/guardian pair will be randomly assigned to either PB no-added-fat, AHA or MED.

DETAILED DESCRIPTION:
Background: There is a need to have effective lifestyle modifications that target the growing group of obese children with dyslipidemia. The beneficial health effects of plant-based (PB) diets in adults are known. Studies have suggested that a low-fat vegan diet (no animal products) may promote weight loss, lower body mass index (BMI), and improve lipoprotein profiles and insulin sensitivity and possibly prevent cardiovascular disease (CVD).1-5 Those who follow a vegetarian diet(no animal products except for dairy and/or eggs) typically have lower cholesterol levels and a lower risk for heart disease than non-vegetarians.6-8 Additionally, vegetarian diets have been shown to not only prevent but reverse heart disease in adults.9-11 The three major diets emphasized in the 2015 United States Dietary Guidelines are a Plant-based Diet (PB), and the American Heart Association-like Diet (AHA) and Mediterranean Diet (MED).(11) Similar to the PB, the AHA diet encourage fruits, vegetables, whole grains, and low sodium intake but permits non-whole grains, low-fat dairy, selected plant oils, and lean meat and fish in moderation. The MED, is similar to AHA with more emphasis on fish and extra virgin olive oil and/or nuts).

Study Aims: The primary aim of this study is to determine whether a PB and/or AHA and/or MED diets significantly change anthropometric measurements and/or biomarkers of CVD risk after a 4 and 52-week intervention in obese children with hypercholesterolemia ages 9-18 years and one of their parents. The investigators also aim to prospectively determine for the first time in children and adults if there are significant outcome differences between the three diets highlighted in the 2015 U.S. Dietary Guidelines.

Protocol Summary The purpose of this research is to investigate the effects of a PB no- added-fat and the AHA and MED in obese (BMI >95%) children ages 9-18 with hypercholesterolemia (>169 mg/dl) and a parent or guardian. Eligible patients will be identified by utilizing the Pediatric Obesity Registry. When possible, in-person discussions or phone calls with their primary or tertiary care physicians will introduce eligible patients and their parents to the study. All eligible patients and parents will receive letters describing the study and requesting their participation. Subjects can choose not to participate in the study, and their health care will not be affected in any way. Subjects not participating will be asked if they are willing to answer a brief questionnaire about why they chose not to participate. The proposed study will be carried out for a total of 52 weeks. The investigators expect to recruit a total of 180 participants (30 children and 30 parents/guardians in each of the three groups). Each child and parent/guardian pair will be randomly assigned to either PB no-added-fat, AHA or MED.

Procedures of the study:

Eligible patients and parent/guardian pairs who are interested in participating in the study will have an initial phone call with the study team to answer any questions regarding the study. Informed consent, or assent for children under age 18, will then be obtained by study team investigators face-to-face with the parent/guardian and child pairs prior to the start of the study at a mutually convenient time and place at Cleveland Clinic Regional and Main Campus sites. Patient and parent/guardian pairs will be randomized to one of the three diets at the first study visit.

Throughout the 52 week diet study, participants will be asked to attend group sessions held on Saturdays during weeks 0, 1, 2, 3, 4, and 52 to learn about their assigned diets and receive support for their efforts. There will Saturday support sessions during weeks 6, 10, 16, 24, 34, and 46 and support phone calls every 2 weeks.

The participants will also provide 24 hour dietary recalls of 2 weekdays and 1 weekend day on three time points: before the first study visit, between weeks 2 and 4, and then between weeks 48 and 52.

Participants will have fasting blood tests to assess biomarkers of cardiovascular risk and anthropometric measurements will be performed weeks 0, 4, and 52. Stool and urine specimens will be obtained for possible future testing for microbiome, genomic data and markers of cardiovascular risk at weeks 0, 4, and 52.

ELIGIBILITY:
Inclusion Criteria:

* children ages 9-18
* obese (BMI >95%)
* hypercholesterolemia (>169 mg/dl)

Exclusion Criteria:

* pregnant women

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline Biomarkers of Cardiovascular Risk at 4 weeks and 52 weeks | baseline, 4 weeks, 52 weeks
  Change in lipid panel, myeloperoxidase, hs C-reactive protein, insulin, glucose, HgbA1C, ALT, AST levels at 4 weeks and 52 weeks after baseline

SECONDARY OUTCOMES:
Change from baseline weight at 4 weeks and 52 weeks | baseline, 4 weeks, 52 weeks
  Change in kilograms at 4 weeks and 52 weeks after baseline
Change from baseline blood pressure at 4 weeks and 52 weeks | baseline, 4 weeks, 52 weeks
  Change in systolic blood pressure in mm Hg at 4 weeks and 52 weeks after baseline
Change in baseline waist circumference at 4 weeks and 52 weeks | baseline, 4 weeks, 52 weeks
  Change in centimeters at 4 weeks and 52 weeks after baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnard ND, Cohen J, Jenkins DJ, Turner-McGrievy G, Gloede L, Jaster B, Seidl K, Green AA, Talpers S. A low-fat vegan diet improves glycemic control and cardiovascular risk factors in a randomized clinical trial in individuals with type 2 diabetes. Diabetes Care. 2006 Aug;29(8):1777-83. doi: 10.2337/dc06-0606. PMID 16873779
- [Background] Barnard ND, Scialli AR, Turner-McGrievy G, Lanou AJ, Glass J. The effects of a low-fat, plant-based dietary intervention on body weight, metabolism, and insulin sensitivity. Am J Med. 2005 Sep;118(9):991-7. doi: 10.1016/j.amjmed.2005.03.039. PMID 16164885
- [Background] Ferdowsian HR, Barnard ND. Effects of plant-based diets on plasma lipids. Am J Cardiol. 2009 Oct 1;104(7):947-56. doi: 10.1016/j.amjcard.2009.05.032. PMID 19766762
- [Background] Mishra S, Xu J, Agarwal U, Gonzales J, Levin S, Barnard ND. A multicenter randomized controlled trial of a plant-based nutrition program to reduce body weight and cardiovascular risk in the corporate setting: the GEICO study. Eur J Clin Nutr. 2013 Jul;67(7):718-24. doi: 10.1038/ejcn.2013.92. Epub 2013 May 22. PMID 23695207
- [Background] Turner-McGrievy GM, Barnard ND, Scialli AR. A two-year randomized weight loss trial comparing a vegan diet to a more moderate low-fat diet. Obesity (Silver Spring). 2007 Sep;15(9):2276-81. doi: 10.1038/oby.2007.270. PMID 17890496
- [Background] Fraser GE. Vegetarian diets: what do we know of their effects on common chronic diseases? Am J Clin Nutr. 2009 May;89(5):1607S-1612S. doi: 10.3945/ajcn.2009.26736K. Epub 2009 Mar 25. PMID 19321569
- [Background] Hu FB. Plant-based foods and prevention of cardiovascular disease: an overview. Am J Clin Nutr. 2003 Sep;78(3 Suppl):544S-551S. doi: 10.1093/ajcn/78.3.544S. PMID 12936948
- [Background] Tuso PJ, Ismail MH, Ha BP, Bartolotto C. Nutritional update for physicians: plant-based diets. Perm J. 2013 Spring;17(2):61-6. doi: 10.7812/TPP/12-085. PMID 23704846
- [Background] Esselstyn CB Jr, Gendy G, Doyle J, Golubic M, Roizen MF. A way to reverse CAD? J Fam Pract. 2014 Jul;63(7):356-364b. PMID 25198208
- [Background] Ornish D, Scherwitz LW, Billings JH, Brown SE, Gould KL, Merritt TA, Sparler S, Armstrong WT, Ports TA, Kirkeeide RL, Hogeboom C, Brand RJ. Intensive lifestyle changes for reversal of coronary heart disease. JAMA. 1998 Dec 16;280(23):2001-7. doi: 10.1001/jama.280.23.2001. PMID 9863851
- [Background] U.S. Department of Health and Human Services and U.S. Department of Agriculture. 2015-2020 Dietary Guidelines for Americans. 8th Edition. December 2015. Available at http://health.gov/dietaryguidelines/2015/guidelines/
- [Background] Macknin M, Kong T, Weier A, Worley S, Tang AS, Alkhouri N, Golubic M. Plant-based, no-added-fat or American Heart Association diets: impact on cardiovascular risk in obese children with hypercholesterolemia and their parents. J Pediatr. 2015 Apr;166(4):953-9.e1-3. doi: 10.1016/j.jpeds.2014.12.058. Epub 2015 Feb 12. PMID 25684089